CLINICAL TRIAL: NCT01743638
Title: Technical Success, Safety, and Short-term Efficacy for MR-Guided Laser Ablation of Prostate Bed Recurrences
Brief Title: MR-Guided Laser Ablation of Prostate Bed Recurrences
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Woodrum, Assistant Professor of Radiology, Mayo Clinic, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-001584
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Prostate Tumors
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MR-Guided Laser Ablation (Experimental)
  Interventions: Procedure: MR-Guided Laser Ablation

INTERVENTIONS:
Procedure: MR-Guided Laser Ablation

SUMMARY:
The purpose of this study is to see if MR-guided laser ablation can effectively treat prostate tumor recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Patients with "biopsy proven" soft tissue tumor recurrences of prostate fossa referred to Urology and/or Interventional Radiology for treatment.
* Surgery is not a desirable alternative therapy at the time of enrollment
* Radiation therapy has failed or not indicated or can be safely postponed
* Tumor size ≤ 5 cm at its largest diameter
* Tumor does not encompass the rectal wall or external urethral sphincter
* Performance status is ECOG 2 or better in adults
* Patient is able to undergo MRI

Exclusion Criteria:

* Patients with pacemaker or defibrillator

Ages: 50 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Measurement of target lesion(s) dimensions at 3-6 month imaging follow-up | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: David A. Woodrum, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States